CLINICAL TRIAL: NCT00564421
Title: A Phase 3 Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple Dose Safety and Efficacy Study of Epinastine Nasal Spray vs. Placebo in Subjects With Seasonal Allergic Rhinitis
Brief Title: Safety and Efficacy Study of Epinastine Nasal Spray in Subjects With Seasonal Allergic Rhinitis (P08648)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P08648; 033-103
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Epinastine low concentration:low dose volume (Experimental)
  Interventions: Drug: epinastine nasal spray, low concentration, low dose volume
- Epinastine low concentration:high dose volume (Experimental)
  Interventions: Drug: epinastine nasal spray, low concentration, high dose volume
- Epinastine high concentration:low dose volume (Experimental)
  Interventions: Drug: epinastine nasal spray, high concentration, low dose volume
- Epinastine high concentration:high dose volume (Experimental)
  Interventions: Drug: epinastine nasal spray, high concentration, high dose volume
- Placebo nasal spray (Placebo Comparator)
  Interventions: Other: placebo nasal spray

INTERVENTIONS:
Drug: epinastine nasal spray, low concentration, low dose volume — 2 sprays in each nostril, dosed twice a day
  Arms: Epinastine low concentration:low dose volume
Other: placebo nasal spray — 2 sprays in each nostril, dosed twice a day
  Other Names: Placebo
  Arms: Placebo nasal spray
Drug: epinastine nasal spray, low concentration, high dose volume — 2 sprays in each nostril, dosed twice a day
  Arms: Epinastine low concentration:high dose volume
Drug: epinastine nasal spray, high concentration, low dose volume — 2 sprays in each nostril, dosed twice a day
  Arms: Epinastine high concentration:low dose volume
Drug: epinastine nasal spray, high concentration, high dose volume — 2 sprays in each nostril, dosed twice a day
  Arms: Epinastine high concentration:high dose volume

SUMMARY:
The purpose of this study is to determine the safety and efficacy of epinastine nasal spray compared to placebo for the treatment of subjects with seasonal allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* A documented history of seasonal allergic rhinitis to mountain cedar or other spring pollen

Exclusion Criteria:

* Significant medical condition
* Significant nasal abnormality
* Significant cardiac condition
* Recent infection
* Use of other allergy medication during the study
* Use of asthma medication other than as-needed albuterol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2007-12-18 (Actual); Primary Completion 2008-02-14 (Actual); Study Completion 2008-02-14 (Actual)

PRIMARY OUTCOMES:
Change in nasal symptom scores | 14 days

SECONDARY OUTCOMES:
Change in ocular symptom scores and quality of life scores | 14 days
Standard safety assessments | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Donald Kellerman, PharmD, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php